CLINICAL TRIAL: NCT01270529
Title: Pedometers to Assess and Increase Physical Activity Among Children With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-03869
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Results first posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Kidney Disease
Keywords: Physical Activity; Physical Performance; Physical Functioning; CKD; ESRD; Transplant Recipients
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Kidney Failure, Chronic

ARMS (3):
- CKD Stages 1-4 (Experimental)
  Interventions: Other: Increasing Physical activity
- ESRD on Dialysis (Experimental)
  Interventions: Other: Increasing Physical activity
- Kidney Transplant recipients (Experimental)
  Interventions: Other: Increasing Physical activity

INTERVENTIONS:
Other: Increasing Physical activity — The subjects (CKD Stages 1-4, ESRD on Hemodialysis or Peritoneal Dialysis) will continue to wear the pedometer for 12 weeks during which time he or she will be asked to gradually increase steps walked per day above baseline physical activity. The patient will be called once a week in order to monitor progress, set new weekly step goals (usually 500-1000 steps/day greater than the previous week), and also to motivate the participant.

SUMMARY:
Hypothesis #1: Most children with CKD stages 2-4, ESRD and kidney transplantation will report participation in physical activity that falls short of recommended levels of physical activity; Children on dialysis will be less active.

Hypothesis #2: Patients will endorse many barriers to physical activity, some of which will be related to their disease or its treatment; those who are less active will endorse more barriers.

Hypothesis #3: Patients will increase their participation in physical activity in response to a pedometer-based 12 week intervention.

Baseline level of physical activity and magnitude of increase in physical activity will be more closely associated with change in physical functioning and performance than stage of kidney disease or type of renal replacement therapy.

Exercise capacity of the child will be measured by the six minute walk test whereby the subject will asked to walk as far as possible in 6 minutes in a straight corridor.

Body fat or body composition will then be measured by Bioelectric Impedance Spectroscopy.

Physical functioning or Health Related Quality of Life will be assessed self reported/ parent proxy reliable and validated questionnaire specifically designed for child with chronic kidney disease called Pediatric Quality of Life Inventory (Peds QL 4.0). Subjects (teens) or parents will also be asked to fill out a questionnaire on barriers to physical activity on their first visit.

Physical activity will be measured in the form of daily steps. The child will wear the pedometer for the first week to assess his/her baseline level of activity. Then the child will continue to wear the pedometer for another 12 weeks during which time he or she will be asked to gradually increase steps walked per day above baseline physical activity. The patient will be called once a week in order to monitor progress, set new weekly step goals (usually 500-1000 steps/day greater than the previous week), and motivate the participant.

After 12 weeks of the pedometer-based intervention to increase physical activity, physical performance, body composition and physical functioning (as described above) will be measured once again to assess the effect of increased physical activity on a second visit.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, male and female, aged 6-20 years.
* Chronic kidney disease stages 2-4 and ESRD on peritoneal dialysis or hemodialysis and kidney transplantation.
* Patients who can follow simple commands.
* English and Spanish speaking only.

Exclusion Criteria:

* Patients hospitalized in the past 1 month.
* Patients hospitalized in the past I month for infection.
* Patients hospitalized in the past 1 month post peritoneal or hemodialysis catheter placement for the first time.
* 1 month after starting renal replacement therapy for the first time.
* 3 months post kidney transplantation.
* In the opinion of the investigator too ill to participate.
* Unwilling to participate.
* Language barrier.
* Patient with any signs of active infection, shortness of breath, trauma or injury to the legs or feet or those undergoing cardiac evaluation.
* Patients unable to verbalize discomfort or developmental delay will not be included.
* Patients with respiratory distress or on oxygen will be excluded.
* Parents or subjects unable to afford transportation for the 2 scheduled visits will also be excluded.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CKD Stages 1-4 | ESRD on Dialysis | Kidney Transplant Recipients
Started | 12 | 7 | 25
Completed | 12 | 7 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CKD Stages 1-4 | ESRD on Dialysis | Kidney Transplant Recipients | Total
Number analyzed (Participants) | 12 | 7 | 25 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (3.6) | 14.7 (2.1) | 14.8 (3.6) | 15.1 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11 | 22
  Male | 5 | 3 | 14 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic white | 4 | 1 | 7 | 12
  Hispanic | 5 | 3 | 12 | 20
  Asian American | 1 | 2 | 5 | 8
  African American | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity
Description: Participants will measure physical activity in the form of daily steps using a pedometer
Time Frame: Baseline, 12 weeks
Measure: Mean (95% Confidence Interval); unit: change in steps per day
Arm/Group | CKD Stages 1-4 | ESRD on Dialysis | Kidney Transplant Recipients
Number analyzed (Participants) | 12 | 7 | 25
change in steps per day | 73 [-115 to 262] | -133 [-325 to 58] | 100 [-14 to 208]

ADVERSE EVENTS:
Arm/Group | CKD Stages 1-4 | ESRD on Dialysis | Kidney Transplant Recipients
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/7 | 0/25
Other Adverse Events (participants affected / at risk) | 0/12 | 0/7 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No